CLINICAL TRIAL: NCT06142799
Title: Post-treatment Pain After Cementing an Indirect Restoration at the End of a Root Canal Treatment: Clinical Trial
Brief Title: Influence of Moment of Restoration in Pain After a Root Canal Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REST-ECL-2023-09
Record Dates: First submitted 2023-11-15; First posted 2023-11-22 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-09

CONDITIONS: Irreversible Pulpitis; Pulp Necroses
Keywords: root canal treatment; cusp coverage
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate overlay placement (Experimental): Immediately after root canal treatment an overlay is cemented, and the patient is asked to record the pain after 6, 12, 24, 48 and 72 hours after treatment
  Interventions: Procedure: root canal treatment
- delayed overlay placement (Active Comparator): After root canal treatment the tooth is left in infraoclussion and the patient is asked to record the pain after 6, 12, 24, 48 and 72 hours
  Interventions: Procedure: root canal treatment

INTERVENTIONS:
Procedure: root canal treatment — The root canal completedwill be completed. Then randomly it will be decided if the planned and milled overlay is placed the same day or delayed one week

SUMMARY:
The goal of this randomized clinical trial is to compare immediate placement of an overlay after root canal treatment with delayed placement of the overlay leaving the tooth one week in infra occlusion. The main question it aims to answer are:

type of study: clinical trial participant population/health conditions: patients more that 18 years old who need a root canal treatment in posterior teeth with antagonist teeth.

question 1: postoperative pain after 6 hours question 2: postoperative pain after 12 hours question 3: postoperative pain after 24 hours question 4: postoperative pain after 48 hours question 4: postoperative pain after 72 hours

If there is a comparison group: Researchers will compare immediate overlay placement and delayed (1 week) overlay placement after root canal treatment to see if there is more pain in one group than in the other.

DETAILED DESCRIPTION:
Introduction: International consensuses on restoration of the root filled teeth recommend early placement of indirect cuspal coverage in posterior teeth. Some classical schools of thought have argued that after endodontic treatment there may be slight periapical inflammation that may lead to over-occlusion, this causing postoperative pain, so that it is preferable to leave the tooth in slight under-occlusion and defer the definitive restoration. Recent studies question this theory and propose a restoration with normal occlusion at the same time of root canal treatment, if possible. Even in these cases, the placement of a full coverage indirect restoration is postponed due to the material impossibility of fabricating it with traditional systems. Modern computer assisted design (CAD)/ computer assisted manufacture (CAM) dental systems make it possible to produce and place such restorations in the same session as the endodontic work is completed. This greatly reduces chair time and the number of visits, while increasing the strength of the tooth right from the start. This is why in this study we compare postoperative pain in two groups of endodontically treated teeth, one in which the indirect CAD/CAM restoration is performed on the same day as the endodontic treatment, and the other in which it is postponed for a week, leaving the tooth in underocclusion.

Background and current status of the subject:

The main reason for root filled teeth loss is restorative failure, which accounts for 60% of all failures. This is followed in order of frequency by periodontal failure, which accounts for 30% of the total. Purely endodontic failure accounts for only 10% of all failures. On the other hand, we know about the high success rate and even higher survival rate of endodontically treated teeth. In a follow-up study of 1462936 endodontic procedures, an 8-year survival rate of 97% was observed. It is accepted that the success, a more demanding criterion than survival, of these root canals ranges between 85 and 90%. Given that most failures occur in the first two years, and given, as already mentioned, that the main cause of this failure is inadequate reconstruction, it has been advised to proceed to definitive restoration of the tooth with an indirect veneering material, and as early as possible.

Modern CAD/CAM systems, and especially the CEREC system, make it possible to produce high-quality chairside indirect restorations in a short time. This makes it possible to place the indirect restoration in a single session. With an appropriate strategy, it is possible to make impressions of the restoration before the root canal treatment is completed. Thus, while the treatment is being completed, the restoration can be fabricated and immediately placed in the tooth without removing the rubber dam isolation at the same visit as the root canal treatment is completed.

After root canal treatment it is possible that periapical inflammation may occur, leading to some overeruption of the tooth. It has been said that this can be a cause of postoperative pain. Thus, there are authors who question the performance of the definitive full-volume restoration on the same day of endodontics, preferring to leave the tooth with a provisional restoration in infraocclusion. However, the literature is not clear regarding a possible increase in postoperative pain in the case of leaving a definitive restoration at full volume, while questioning the relationship between postoperative pain and the type of restoration on the day of endodontics.

In this study, a clinical trial was carried out to compare postoperative pain in endodontically treated teeth in which an indirect restoration of CEREC Tessera was placed on the day of endodontics with another group in which a provisional restoration was left in place and the placement of the restoration with the same material was postponed by one week.

Objectives:

To compare the postoperative pain in endodontically treated teeth with an immediate indirect CAD/CAM restoration after completion of endodontics with that of another group of endodontically treated teeth in which the definitive restoration is deferred for one week.

Working hypothesis:

H0: There is no clinical difference in postoperative pain in patients undergoing endodontics with immediate placement of the definitive restoration and another in which the definitive restoration is deferred for one week.

H1: There is a clinical difference in postoperative pain between patients undergoing endodontic treatment with immediate placement of the definitive restoration and one who defers the definitive restoration for one week.

Material and methods: 30 patients will be recruited for the study. Inclusion criteria: Patients requiring root canal treatment on a molar without acute pain.

Exclusion criteria: Age less than 18 years. An optical impression of the problem arch, the antagonist arch and the intermaxillary relationship will be taken using a Primescan intraoral scanner (software version 5.2.4) according to the manufacturer's recommended protocol. All scans shall be taken by the same operator (J.E.), with four years of routine clinical use of the same device. The tooth shall then be isolated with a rubber dam, covering at least three additional teeth to the problem tooth. Once the dam is in place, the original scan of the problem tooth (control scan) is retrieved and a copy is made and saved as a biocopy. In the biopsy, the problem tooth and the proximal sides of the adjacent teeth shall be trimmed using the cutting tool, taking care to distance the limits of the margins and the proximal contact points.

The tooth is reconstructed, removing the caries if necessary. If the pulp is exposed, the pulp is filled with Teflon prior to restoration of the tooth. Once the composite restoration has been completed, the tooth will be milled for the final restoration that is considered appropriate. Next, the problem tooth will be scanned again, starting from the occlusal surface, to facilitate the virtual coincidence between both scans, and making sure that the margins of the restoration and the proximal faces of the adjacent teeth were well captured (test scan). From these scans, the restoration will be designed and fabricated in Tessera material (Lithium disilicate). While the restoration is being produced, the root canal treatment will be carried out. The canal opening will be made, the location of the canals with K type files and instrumentation with WaveOne files. If necessary, the instrumentation is completed with Profile files. A VDW Gold motor is used for the instrumentation of the canals and the determination of the working length. The canals are thoroughly irrigated with 4% sodium hypochlorite, followed by 96° alcohol, 15% ethylenediaminetetraacetic acid (EDTA) for 30 seconds, then alcohol again, then 4% sodium hypochlorite again and finally alcohol. Once irrigation is complete, the canals are dried with sterile paper tips, and then sealed with Thermafil@ and AH-Plus@ cement. The Thermafil shanks are cut, the excess gutta-percha is removed from the chamber and the cement residues are cleaned with a cotton wool soaked in alcohol.

Once the endodontic treatment has been completed, a random decision is made as to whether a permanent or temporary restoration is to be placed. In case of a temporary restoration, the access is filled with Cavit and the rubber dam is removed. In case of a definitive restoration, the tooth surface is treated for bonding (50micron aluminium oxide blasting, acid etching with 30% orthophosphoric acid, rinsing, drying, priming and bonding). The adhesive surface of the Tessera restoration is etched with 5% hydrofluoric acid for 30 seconds, rinsed with water, etched with 30% orthophosphoric acid for 30 seconds, rinsed, silane bonded for 1 minute and adhesive bonded. The restoration is then cemented with Dual cement, and the rubber dam is removed.

Pain is assessed using a visual analogue scale (VAS) without scales. The patient is given a sheet of paper with a 10 cm line on the outside (left) marked "no pain" and on the outside (right) marked "a lot of pain". The patient is asked to draw a mark on the line in the position that he/she considers corresponds to the pain he/she will experience. The distance from the left end to the patient's mark will be measured and used for pain assessment. Records will be taken at 6 hours, 12 hours, 24 hours, 48 hours and 72 hours. At one week the patient shall return to the practice to return the control sheet and, if necessary, verify the occlusal adjustment or placement of the definitive restoration.

Analysis of results: The sample was calculated by means of G power 3 software version 3.1.9, power 80% and alpha=0.05. The normal distribution and homogeneity of variances of the values of the VAS measurements will be verified by Shapiro-Wilk and Levene tests. Statistical significance of differences in means between test and control groups will be determined by means of parametric tests (Student's t-test).

ELIGIBILITY:
Inclusion Criteria:

* Need of a root canal treatment in a posterior tooth

Exclusion Criteria:

* Preoperative pain requiring pain killers
* Absence of antagonist teeth
* cannot afford and overlay

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | 6, 12, 24, 48, 72 hours
  Pain assessed by the visual analog scale. A 10 cm line with the words "extreme pain" and "no pain" will be used

CONTACTS AND LOCATIONS:
Overall Officials: MARC GARCIA, DDS, PhD, Study Director — Universitat Internacional de Catalunya
Locations (2):
- Spain (2):
  - Clinica Universitaria d'Odontologia, Sant Cugat Del Vallés, Barcelona
  - Clinica Lluch, Barcelona